CLINICAL TRIAL: NCT00135356
Title: A Phase IV, Open-Label, Randomized, Multicenter Trial Assessing a Reyataz-Based Substitution Approach in the Management of Lipodystrophy Syndrome. Research Into Atazanavir in Lipodystrophy (The REAL Study)
Brief Title: Study of Reyataz in HIV-infected Patients With Lipodystrophy Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI424-131
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Results first posted 2010-05-07 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-04

CONDITIONS: HIV-Associated Lipodystrophy Syndrome
Keywords: HIV infections
MeSH Terms: conditions — HIV-Associated Lipodystrophy Syndrome; HIV Infections | interventions — Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Switch arm (Active Comparator)
  Interventions: Drug: Atazanavir (ATV) + ritonavir (RTV), continuation of backbone 2 nucleoside reverse transcriptase inhibitor (NRTIs)
- Control Arm (Active Comparator)
  Interventions: Drug: continuation of current HAART (boosted protease inhibitor [PI] combination + 2 NRTIs)

INTERVENTIONS:
Drug: Atazanavir (ATV) + ritonavir (RTV), continuation of backbone 2 nucleoside reverse transcriptase inhibitor (NRTIs) — Capsules, Oral, ATV 300 mg + RTV 100 mg once daily up to 96 weeks
  Other Names: Reyataz
  Arms: Switch arm
Drug: continuation of current HAART (boosted protease inhibitor [PI] combination + 2 NRTIs) — Protease inhibitor [PI] combination + 2 NRTIs
  Arms: Control Arm

SUMMARY:
The purpose of this clinical research study is to learn if human immunodeficiency virus (HIV)-infected subjects with abdominal fat accumulation on their highly active antiretroviral treatment (HAART) regimen have better changes in fat distribution after switching to atazanavir-ritonavir than those remaining on their current protease inhibitor boosted HAART regimen.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected on HAART regimen containing 2 NRTI and boosted PI for at least 12 weeks prior to screening. Subjects may not have experienced virological failure to more than one prior PI-containing regimen. Must be able to swallow tablets
* Viral load <400 c/mL at screening and stable for at least 6 months
* Signs of fat redistribution and lipohypertrophy (abdominal) Waist to Hip Ratio >0.90 and Waist Circumference >88.2 cm for men and Waist Circumference >75.3 for women

Exclusion Criteria:

* Pregnant or breastfeeding women
* New HIV-related opportunistic infections
* Active alcohol or substance use
* Grade 4 lab toxicity
* History of taking atazanavir (ATV)
* Prohibited therapies, including non-nucleoside reverse transcriptase inhibitors (NNRTI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2005-07; Primary Completion 2007-07 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (30):
- United States (4):
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Honolulu, Hawaii
  - Local Institution, Huntersville, North Carolina
  - Local Institution, Houston, Texas
- Canada (2):
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
- France (5):
  - Local Institution, Bondy
  - Local Institution, Lagny-sur-Marne
  - Local Institution, Lyon
  - Local Institution, Nice
  - Local Institution, Paris
- Germany (2):
  - Local Institution, Frankfurt am Main
  - Local Institution, München
- Italy (4):
  - Local Institution, Brescia
  - Local Institution, Milan
  - Local Institution, Modena
  - Local Institution, Roma
- Mexico (3):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Puebla City
- Poland (2):
  - Local Institution, Szczecin
  - Local Institution, Wroclaw
- Spain (6):
  - Local Institution, Barcelona
  - Local Institution, Elche (Alicante)
  - Local Institution, Guipuzcoa
  - Local Institution, Madrid
  - Local Institution, Málaga
  - Local Institution, Valencia
- United Kingdom (2):
  - Local Institution, Brighton, East Sussex
  - Local Institution, London, Greater London

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 219 participants were enrolled and 18 were never randomized (1 poor/noncompliance; 10 no longer met study criteria; 5 withdrew consent). 201 participants were randomized; however, 1 participant was never treated and is not included in the participant flow.
Groups:
- ATV/RTV Switch Arm: Participants switching their current treatment with a ritonavir (RTV)-boosted protease inhibitor (PI)-containing highly active antiretroviral therapy (HAART) regimen to atazanavir (ATV)/RTV (ATV: 2 x 150 mg capsules once daily (QD) / RTV: 1 x 100 mg capsule QD) while continuing their background nucleoside reverse transcriptase inhibitors (NRTIs).
- PI/RTV Control Arm: Participants continued on their current treatment with an RTV-boosted, PI-containing HAART regimen while continuing their background NRTIs.
Period: Overall Study
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Started | 131 (Number randomized and treated) | 69 (Number randomized and treated(1 randomized and never treated subject not included in this number.))
Discontinued Prior to Week 96 Visit | 16 | 9
Discontinued on or After Week 96 Visit | 1 | 0
Completed | 114 | 60
Not Completed | 17 | 9
Not completed — Adverse Event | 6 | 2
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Surgery for abdominal fat | 1 | 0
Not completed — Change in antiviral regimen | 0 | 1
Not completed — Poor/noncompliance | 1 | 1
Not completed — No longer meets study criteria | 2 | 0
Not completed — Withdrawal by Subject | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm | Total
Number analyzed (Participants) | 131 | 69 | 200
Age Continuous [Median (Full Range); unit: Years] | 43 [23 to 79] | 42 [26 to 65] | 43 [23 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 14 | 49
  Male | 96 | 55 | 151
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 83 | 43 | 126
  Mestizo | 31 | 15 | 46
  Black/African American | 15 | 10 | 25
  American Indian/Alaska Native | 1 | 0 | 1
  Latino/Hispanic | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Europe | 77 | 39 | 116
  North America | 54 | 30 | 84
Cluster of Differentiation 4 (CD4) Distribution [Number; unit: Participants] — CD4=a protein marker on the surface of certain types of T lymphocytes and other cells; HIV binds to CD4 receptors to enter host cells.
  Participants
    50 to <100 cells/mm3 | 2 | 0 | 2
    100 to <200 cells/mm3 | 14 | 3 | 17
    200 to <350 cells/mm3 | 24 | 22 | 46
    350 to <500 cells/mm3 | 31 | 16 | 47
    ≥500 cells/mm3 | 60 | 27 | 87
    Missing | 0 | 1 | 1
Fasting Glucose [Number; unit: participants] — 7 participants in ATV/RTV arm and 3 participants in PI/RTV arm were missing this baseline measurement.
  participants
    <100 mg/dL | 96 [83.0 to 99.0] | 49 [82.0 to 100.0] | 145
    100 mg/dL to <126 mg/dL | 23 | 13 | 36
    >=126 mg/dL | 5 | 4 | 9
Fasting Lipids [Number; unit: participants] — Triglycerides, non-high density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol, total cholesterol, and HDL cholesterol. Values for all baseline fasting lipid measurements were missing for 8 participants in the ATV/RTV arm. Values for baseline fasting LDL cholesterol were missing for 8 participants in the PI/RTV arm; values for all other baseline lipid measurements were missing for 7 participants.
  participants
    Triglycerides <150 mg/dL | 29 [41 to 54] | 14 [35 to 53] | 43
    Triglycerides 150 mg/dL to <200 mg/dL | 28 [139 to 198] | 9 [126 to 192] | 37
    Triglycerides 200 mg/dL to <500 mg/dL | 52 [90 to 143] | 27 [84 to 125] | 79
    Triglycerides >=500 mg/dL | 14 [151 to 326] | 12 [154 to 425] | 26
    Non-HDL Cholesterol <130 mg/dL | 22 [80 to 111] | 16 [78 to 111] | 38
    Non-HDL Cholesterol 130 mg/dL to <160 mg/dL | 31 | 14 | 45
    Non-HDL Cholesterol 160 mg/dL to <190 mg/dL | 32 | 15 | 47
    Non-HDL Cholesterol 190 mg/dL to <220 mg/dL | 22 | 9 | 31
    Non-HDL Cholesterol >=220 mg/dL | 16 | 8 | 24
    LDL Cholesterol <100 mg/dL | 40 | 22 | 62
    LDL Cholesterol 100 mg/dL to <130 mg/dL | 36 | 25 | 61
    LDL Cholesterol 130 mg/dL to <160 mg/dL | 30 | 11 | 41
    LDL Cholesterol 160 mg/dL to <190 mg/dL | 11 | 1 | 12
    LDL Cholesterol >=190 mg/dL | 6 | 2 | 8
    Total Cholesterol <200 mg/dL | 45 | 28 | 73
    Total Cholesterol 200 mg/dL to 240 mg/dL | 42 | 19 | 61
    Total Cholesterol 240 mg/dL to 300 mg/dL | 29 | 11 | 40
    Total Cholesterol >=300 mg/dL | 7 | 4 | 11
    HDL Cholesterol <40 mg/dL | 23 | 21 | 44
    HDL Cholesterol 40 mg/dL to <60 mg/dL | 80 | 32 | 112
    HDL Cholesterol >=60 mg/dL | 20 | 9 | 29
Human Immunodeficiency Virus Ribonucleic Acid (HIV RNA) Distribution [Number; unit: Participants]
  <50 c/mL | 117 | 64 | 181
  50 to <400 c/mL | 10 | 5 | 15
  400 to <1000 c/mL | 2 | 0 | 2
  ≥1000 c/mL | 2 | 0 | 2
Adipose Tissue at Baseline [Median (Inter-Quartile Range); unit: cm2] — Visceral, subcutaneous, and total adipose tissue (VAT, SAT, and TAT) as assessed by computed tomography (CT). Values for all 3 measurements were missing for 20 participants in the ATV/RTV arm (n=111). Values for all 3 measurements were missing for 10 participants in the PI/RTV arm (n=59).
  cm2
    VAT | 131.9 [93.8 to 185.8] | 128.1 [95.8 to 193.7] | 129.4 [94.3 to 186.1]
    SAT | 209.5 [123.6 to 300.7] | 183.9 [151.4 to 282.4] | 193.6 [140.3 to 289.2]
    TAT | 356.2 [263.9 to 446.3] | 328.6 [287.3 to 457.8] | 352.0 [268.5 to 453.1]
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m2] — 131 participants in ATV/RTV arm and 67 participants in PI/RTV arm had this baseline measurement.
  kg/m2 | 25.9 [24.1 to 28.5] | 25.7 [24.2 to 28.8] | 25.9 [24.2 to 28.5]
Body Weight [Median (Inter-Quartile Range); unit: kg] | 75 [69 to 83] | 77 [69 to 87] | 76 [69 to 84]
CD4 Cell Count [Median (Full Range); unit: cells/mm3] — CD4 cell=a type of white blood cell that bears the CD4 surface receptor and helps coordinate a range of immune system activities.
  cells/mm3 | 470 [90 to 1919] | 437 [100 to 1078] | 459 [90 to 1919]
Trunk Fat, Limb Fat, Total Body Fat [Median (Inter-Quartile Range); unit: kg] — Values for all 3 baseline fat measurements were missing for 14 participants in the ATV/RTV arm (n=117). Values for baseline trunk fat measurements were missing for 10 participants in the PI/RTV arm (n=59); values for baseline limb fat and total body fat measurements were missing for 13 participants in the PI/RTV arm (n=56).
  kg
    Trunk Fat | 11.8 [8.6 to 15.3] | 10.9 [8.8 to 13.8] | 11.4 [8.7 to 14.6]
    Limb Fat | 7.1 [4.6 to 10.4] | 6.7 [4.6 to 9.4] | 7.0 [4.6 to 10.0]
    Total Body Fat | 20.8 [14.1 to 26.0] | 18.7 [15.6 to 22.4] | 19.8 [14.8 to 25.7]
Trunk-to-Limb Fat Ratio [Median (Inter-Quartile Range); unit: ratio] — 117 participants in ATV/RTV arm and 56 participants in PI/RTV arm had this measure at baseline.
  ratio | 1.59 [1.27 to 2.04] | 1.73 [1.17 to 2.15] | 1.62 [1.23 to 2.10]
Waist Circumference [Median (Inter-Quartile Range); unit: cm] | 94 [90 to 103] | 95 [91 to 100] | 94 [90 to 102]
Waist-to-Hip Ratio [Median (Inter-Quartile Range); unit: ratio] — 131 participants in ATV/RTV arm and 68 participants in PI/RTV arm had this baseline measurement.
  ratio | 0.99 [0.95 to 1.03] | 0.97 [0.94 to 1.02] | 0.99 [0.95 to 1.03]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trunk-to-limb Fat Ratio as Measured by Dual Energy X-Ray Absortiometry (DEXA) at Week 48
Description: Mean changes from Baseline in trunk-to-limb fat ratio as measured by DEXA, an x-ray scan used to measure bone mineral density. Clinical improvement is associated with a decrease in values. (Baseline trunk-to-limb fat ratio values can be found in the Baseline Characteristics section.)
Time Frame: Baseline, Week 48
Population: Treated participants. Observed case (OC) analysis: n=participants with fat measurement at baseline and at the analysis timepoint. Last observation carried forward (LOCF): n=participants with fat measurement at baseline and at or before the analysis timepoint.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 131 | 69
ratio
  LOCF Population (n=112; n=54) | 0.02 (0.027) | -0.02 (0.036)
  OCPopulation (n=105; n=51) | 0.02 (0.029) | -0.01 (0.038)
Statistical Analysis 1: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; LOCF; Test type: Superiority or Other; p = 0.48, t-test, 2 sided — P-value not adjusted for multiple testing, 2-sided 95% CI; Difference in Means = 0.03, 95% CI [-0.06 to 0.12]
Statistical Analysis 2: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; OC; Test type: Superiority or Other; p = 0.57, t-test, 2 sided — P-value not adjusted for multiple testing. 2-sided 95% CI; Difference in Means = 0.07, 95% CI [-0.07 to 12.0]

2. Secondary Outcome: Change From Baseline in Trunk-to-limb Fat Ratio as Measured by DEXA at Week 96
Description: Mean changes from baseline in trunk-to-limb fat ratio as measured by DEXA, an x-ray scan used to measure bone mineral density. Clinical improvement is associated with a decrease in values.(Baseline trunk-to-limb fat ratio values can be found in the Baseline Characteristics section.)
Time Frame: Baseline, Week 96
Population: Observed case (OC) analysis: n=participants with fat measurement at baseline and at the analysis timepoint. Last observation carried forward (LOCF): n=participants with fat measurement at baseline and at or before the analysis timepoint.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 131 | 69
ratio
  LOCF Population (n=112; n=54) | 0.04 (0.035) | 0.02 (0.046)
  OC Population (n=94; n=45) | 0.04 (0.041) | 0.05 (0.051)
Statistical Analysis 1: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; LOCF; Test type: Superiority or Other; p = 0.73, t-test, 2 sided — P-value not adjusted for multiple testing, 2-sided 95% CI; Difference in Means = 0.02, 95% CI [-0.10 to 0.14]
Statistical Analysis 2: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; OC; Test type: Superiority or Other; p = 0.91, t-test, 2 sided — P-value not adjusted for multiple testing, 2-sided 95% CI; Difference in Means = -0.01, 95% CI [-0.14 to 0.13]

3. Secondary Outcome: Mean Percent Change From Baseline in Visceral Adipose Tissue (VAT) Area by Computed Tomography (CT) Scans and in Trunk Fat by DEXA.
Description: The mean percent change from baseline in physical signs of lipohypertrophy, as assessed objectively by changes in visceral adipose tissue (VAT) area (cm2) by computed tomography (CT) scans and by changes in trunk fat (kg) by DEXA. Clinical improvement is associated with a decrease in values. (Baseline values can be found in the Baseline Characteristics section.)
Time Frame: Baseline, Week 48, Week 96
Population: VAT analysis population=treated subjects with adipose tissue pairs (LOCF); trunk fat analysis population=treated subjects with fat pairs (LOCF); n=number of subjects with measurement at baseline and at or before the analysis timepoint.
Measure: Mean (Inter-Quartile Range); unit: Percent change
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 131 | 69
Percent change
  Week 48 VAT (n=98; n=53) | 6.5 [-13.8 to 25.7] | -0.4 [-10.8 to 14.6]
  Week 96 VAT (n=101; n=53) | 4.3 [-11.7 to 26.5] | 2.1 [-12.4 to 23.3]
  Week 48 Trunk Fat (n=112; n=57) | 2.6 [-5.8 to 12.4] | -1.8 [-10.0 to 9.2]
  Week 96 Trunk Fat (n=112; n=57) | 1.6 [-6.7 to 14.3] | -3.6 [-12.9 to 9.5]
Statistical Analysis 1: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; Week 48 VAT LOCF; Test type: Superiority or Other; p = 0.27, t-test, 2 sided — P-value not adjusted for multiple testing, 2-sided 95% CI; Difference in Mean = 5.2, 95% CI [-3.9 to 15.1]
Statistical Analysis 2: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; VAT, Week 96 LOCF; Test type: Superiority or Other; p = 0.68, t-test, 2 sided — P-value not adjusted for multiple testing, 2-sided 95% CI; Difference in Mean = 1.8, 95% CI [-6.7 to 11.2]
Statistical Analysis 3: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; Week 48 Trunk Fat LOCF; Test type: Superiority or Other; p = 0.14, t-test, 2 sided — P-value not adjusted for multiple testing, 2-sided 95% CI; Difference in Means = 4.4, 95% CI [-1.4 to 10.6]
Statistical Analysis 4: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; Week 96 Trunk Fat LOCF; Test type: Superiority or Other; p = 0.14, t-test, 2 sided — P-value not adjusted for multiple testing, 2-sided 95% CI; Difference in Means = 5.3, 95% CI [-1.7 to 12.9]

4. Secondary Outcome: Mean Percent Change From Baseline in Peripheral Adipose Tissue (Limb Fat) by DEXA and by Changes in Subcutaneous Adipose Tissue (SAT) Area by CT Scans
Description: The mean percent change from baseline in physical signs of lipoatrophy, as assessed objectively by changes in peripheral adipose tissue (ie, limb fat (kg) by DEXA and in subcutaneous adipose tissue (SAT) area by CT scans. Clinical improvement is associated with stable values, or an increase in values. (Baseline values can be found in the Baseline Characteristics section.)
Time Frame: Baseline, Week 48, Week 96
Population: SAT analysis population=treated subjects with adipose tissue pairs (LOCF); trunk fat analysis population=treated subjects with fat pairs (LOCF); n=number of subjects with measurement at baseline and at or before analysis timepoint.
Measure: Mean (Inter-Quartile Range); unit: percent change
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 131 | 69
percent change
  Week 48 SAT (n=108; n=59) | -2.2 [-11.6 to 8.7] | -5.9 [-14.4 to 5.8]
  Week 96 SAT (n=111; n=59) | -3.5 [-15.7 to 8.7] | -9.7 [-21.6 to 6.6]
  Week 48 Limb Fat (n=112; 54) | 0.9 [-7.4 to 10.5] | -3.6 [-15.5 to 7.5]
  Week 48 Limb Fat (n=112; n=54) | -0.8 [-11.3 to 12.2] | -6.1 [-19.8 to 8.7]
Statistical Analysis 1: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; SAT, Week 48, LOCF; Test type: Superiority or Other; p = 0.16, t-test, 2 sided — P-value not adjusted for multiple testing, 2-sided 95% CI; Difference in Means = 4.0, 95% CI [-1.6 to 10.0]
Statistical Analysis 2: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; Week 96 SAT; Test type: Superiority or Other; p = 0.06, t-test, 2 sided — P-value not adjusted for multiple testing, 2-sided 95% CI; Difference in Mean = 6.8, 95% CI [-0.2 to 14.2]
Statistical Analysis 3: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; Week 48, Limb Fat; Test type: Superiority or Other; p = 0.15, t-test, 2 sided — P-value not adjusted for multiple testing, 2-sided 95% CI; Difference in Means = 4.6, 95% CI [-1.7 to 11.4]
Statistical Analysis 4: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; Week 96, Limb Fat; Test type: Superiority or Other; p = 0.17, t-test, 2 sided — P-value not adjusted for multiple testing, 2-sided 95% CI; Difference in Means = 5.7, 95% CI [-2.3 to 14.4]

5. Secondary Outcome: Mean Percent Change From Baseline in Total Body Fat by DEXA and in Total Adipose Tissue (TAT) Area by CT Scans
Description: The mean percent change from baseline in total body fat by DEXA and in total adipose tissue (TAT) area by CT scans. Total body fat and TAT are both associated many factors (trunk fat + limb fat + other [weight, etc]), and thus clinical improvement cannot be predicted based solely an increase or decrease of these values. (Baseline values can be found in the Baseline Characteristics section.)
Time Frame: Baseline, Week 48, Week 96
Population: TAT analysis population=treated subjects with adipose tissue pairs (LOCF); trunk fat analysis population=treated subjects with fat pairs (LOCF); n=number of subjects with measurement at baseline and at or before the analysis timepoint
Measure: Mean (Inter-Quartile Range); unit: percent change
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 131 | 69
percent change
  Week 48 TAT (n=108; n= 59) | 0.0 [-9.0 to 10.8] | -3.5 [-12.7 to 10.0]
  Week 96 TAT (n=111; n=59) | -0.9 [-9.2 to 12.7] | -5.0 [-16.0 to 10.4]
  Week 48 Total Body Fat (n=105; n=51) | 1.9 [-5.4 to 11.5] | -3.7 [-10.9 to 5.1]
  Week 96 Total Body Fat (n=94; n=45) | 0.5 [-9.5 to 11.8] | -7.4 [-16.9 to 6.6]
Statistical Analysis 1: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; Week 48 TAT; Test type: Superiority or Other; p = 0.19, t-test, 2 sided — P-value not adjusted for multiple testing, 2-sided 95% CI; DIfference in Means = 3.6, 95% CI [-1.8 to 9.4]
Statistical Analysis 2: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; Week 96 TAT; Test type: Superiority or Other; p = 0.16, Wilcoxon (Mann-Whitney) — P-value not adjusted for multiple testing, 2-sided 95% CI; DIfference in Means = 4.3, 95% CI [-1.7 to 10.7]
Statistical Analysis 3: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; Week 48 Total Body Fat; Test type: Superiority or Other; p = 0.0385, t-test, 2 sided — P-value not adjusted for multiple testing, 2-sided 95% CI; Difference in Means = 5.0, 95% CI [0.3 to 9.7]
Statistical Analysis 4: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; Week 96 Total Body Fat; Test type: Superiority or Other; p = 0.10, t-test, 2 sided — P-value not adjusted for multiple testing, 2-sided 95% CI; Difference in Means = 5.9, 95% CI [-1.0 to 13.2]

6. Secondary Outcome: Mean Percent Changes From Baseline in Fasting Lipids
Description: Mean percent changes from baseline in fasting total, low-density lipoprotein (LDL), high-density lipoprotein (HDL), and non-HDL cholesterol, triglycerides, and apolipoprotein B
Time Frame: Baseline, Week 48, Week 96
Population: Treated Subjects (LOCF). n=56 for LDL cholesterol in the PI/RTV arm at both timepoints
Measure: Number; unit: Percent change
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 122 | 57
Percent change
  Week 48 - Total Cholesterol | -13.0 | -1.0
  Week 48 - HDL Cholesterol | -6.2 | -2.6
  Week 48 - Non-HDL Cholesterol | -14.8 | -0.6
  Week 48 - LDL Cholesterol | -10.4 | 2.6
  Week 48 - Triglycerides | -23.8 | -11.7
  Week 48 - Apolipoprotein B | -7.6 | 1.1
  Week 96 - Total Cholesterol | -12.5 | -0.1
  Week 96 - HDL Cholesterol | -6.8 | -4.6
  Week 96 - Non-HDL Cholesterol | -14.0 | 1.2
  Week 96 - LDL Cholesterol | -8.4 | 3.6
  Week 96 - Triglycerides | -25.0 | -12.2
  Week 96 - Apolipoprotein B | -8.3 | 8.3

7. Secondary Outcome: Mean Changes From Baseline in Fasting Glucose at Week 48 and Week 96
Time Frame: Baseline, Week 48, Week 96
Population: Treated participants (LOCF); n=number of participants with baseline value at or before analysis timepoint.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 131 | 69
mg/dL
  Week 48 (n=124; n=63) | 3.6 (2.60) | -3.3 (2.92)
  Week 96 (n=124; n=64) | 1.2 (2.82) | 3.0 (2.88)

8. Secondary Outcome: Mean Changes From Baseline in Fasting Insulin at Week 48 and Week 96
Time Frame: Baseline, Week 48, Week 96
Population: Treated participants (LOCF); n=number of participants with baseline value at or before analysis timepoint.
Measure: Mean (Standard Error); unit: microunits per milliliter
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 131 | 69
microunits per milliliter
  Baseline (n=124; n=62) | 14.1 (1.04) | 21.8 (3.36)
  Week 48 (n=124; n=59) | 1.3 (1.46) | -4.1 (3.79)
  Week 96 (n=124; n=59) | 0.0 (1.20) | 0.3 (4.76)

9. Secondary Outcome: Mean Changes From Baseline in Fasting Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: HOMA-IR is an index used in evaluation of obese patients at risk for type 2 diabetes which requires fasting glucose and insulin concentrations. It is a mathematical model based on the theory of a negative feedback loop between the liver and β-cells that regulates both fasting glucose and insulin concentrations and can be used to estimate pancreatic β-cell function and degree of insulin resistance. HOMA-IR normal values are between 2 and 2.5. HOMA-IR ≥ 2.5 indicates insulin-resistance.
Time Frame: Baseline, Week 48, Week 96
Population: Treated participants (LOCF); n=number of participants with baseline value at or before analysis timepoint.
Measure: Mean (Standard Error); unit: mg/dL x uU/mL
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 131 | 69
mg/dL x uU/mL
  Baseline (n=115; n=59) | 3.42 (0.309) | 5.43 (1.233)
  Week 48 (n=115; n=57) | 0.74 (0.589) | -1.73 (1.223)
  Week 96 (n=115; n=57) | 0.28 (0.500) | 1.00 (1.648)

10. Secondary Outcome: Mean Changes From Baseline in Body Weight at Week 48 and Week 96
Time Frame: Baseline, Week 48, Week 96
Population: LOCF; n=number of participants with baseline value and value at or before analysis timepoint
Measure: Mean (Standard Error); unit: kg
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 130 | 68
kg
  Week 48 (n=130; n=68) | 1 (0.3) | -1 (0.4)
  Week 96 (n=130; n=68) | 0 (0.4) | -1 (0.7)

11. Secondary Outcome: Mean Changes From Baseline in Waist Circumference at Week 48 and Week 96
Time Frame: Baseline, Week 48, Week 96
Population: LOCF; n=number of participants with baseline value and value at or before analysis timepoint
Measure: Mean (Standard Error); unit: cm
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 131 | 69
cm
  Week 48 (n=123; n=66) | -1 (0.5) | -1 (0.6)
  Week 96 (n=124; n=66) | -1 (0.6) | -1 (0.8)

12. Secondary Outcome: Mean Changes From Baseline in Body Mass Index at Week 48 and Week 96
Time Frame: Baseline, Week 48, Week 96
Population: LOCF; n=number of participants with baseline value and value at or before analysis timepoint
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 131 | 69
kg/m2
  Week 48 (n=130; n=67) | 0.3 (0.12) | -0.2 (0.13)
  Week 96 (n=130; n=67) | 0.2 (0.13) | -0.5 (0.25)

13. Secondary Outcome: Mean Changes From Baseline in Waist-to-Hip Ratio at Week 48 and Week 96
Description: Mean changes from baseline in proportion of waist to hip measurements.
Time Frame: Baseline, Week 48, Week 96
Population: LOCF; n=number of participants with baseline value and value at or before analysis timepoint
Measure: Mean (Standard Error); unit: ratio
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 131 | 69
ratio
  Week 48 (n=123; n=65) | -0.01 (0.005) | -0.01 (0.007)
  Week 96 (n=124; n=65) | -0.01 (0.006) | -0.01 (0.007)

14. Secondary Outcome: Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths, and AEs Leading to Discontinuation
Description: Percentage of Participants with AEs, Serious AEs (SAEs), Deaths, and AEs leading to discontinuation. An AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition. An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a cancer, is a congenital anomaly/birth defect, results in the development of drug dependency or drug abuse, is an important medical event.
Time Frame: Through Week 96 of study therapy
Population: Treated participants
Measure: Number; unit: Percentage of Participants
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 131 | 69
Percentage of Participants
  Death | 0 | 0
  SAE | 8 | 7
  AE Leading to Discontinuation | 5 | 3
  Any AEs (all grades) through Week 96 | 90 | 83

15. Secondary Outcome: Percentage of Participants With Abnormal Liver Function Tests
Description: Percentage of participants with Abnormal Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), and Total Bilirubin (TBILI) measurements. Values for liver tests are graded using the modified World Health Organization (WHO) criteria. Grade 1 is mild, grade 2 is moderate, grade 3 is severe, grade 4 is life threatening or disabling.
Time Frame: Week 48, Week 96
Population: All treated participants
Measure: Number; unit: Percentage of Participants
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 131 | 69
Percentage of Participants
  Wk 48 ALT Grades 1-4 | 34 | 23
  Wk 48 ALT Grades 3-4 | 1 | 0
  Wk 48 ALT Grade 4 | 0 | 0
  Wk 96 ALT Grades 1-4 | 37 | 32
  Wk 96 ALT Grades 3-4 | 2 | 0
  Wk 96 ALT Grade 4 | 0 | 0
  Wk 48 AST Grade 1-4 | 19 | 15
  Wk 48 AST Grades 3-4 | 1 | 0
  Wk 48 AST Grade 4 | 0 | 0
  Wk 96 AST Grades 1-4 | 24 | 19
  Wk 96 AST Grades 3-4 | 1 | 0
  Wk 96 AST Grade 4 | 0 | 0
  Wk 48 TBILI Grades 1-4 | 94 | 19
  Wk 48 TBILI Grades 3-4 | 53 | 0
  Wk 48 TBILI Grade 4 | 13 | 0
  Wk 96 TBILI Grades 1-4 | 95 | 21
  Wk 96 TBILI Grades 3-4 | 60 | 0
  Wk 96 TBILI Grade 4 | 17 | 0

16. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) Leading to Discontinuation
Description: Percentage of Participants with AEs leading to discontinuation of study therapy. An AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition. All events listed in this table were SAEs, except for renal impairment and hypertriglycerideamia, which were an AEs (and did not meet the 5 percent threshold reported in Adverse Event module of this record).
Time Frame: Through Week 96
Population: Treated subjects
Measure: Number; unit: Percent of Participants
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 131 | 69
Percent of Participants
  Any adverse experience leading to discontinuation | 5 | 3
  Hyperbilirubinemia | 2 | 0
  Jaundice | 1 | 0
  Drug abuse | 1 | 0
  Renal impairment | 1 | 0
  Stevens-Johnson syndrome | 1 | 0
  Hypertriglyceridemia | 0 | 1
  Squamous cell carcinoma | 0 | 1

17. Secondary Outcome: Kaplan-Meier Cumulative Proportion of Participants Without Virologic Rebound (HIV RNA ≥400 c/mL) at Timepoints up to Week 96 in Treated Participants With HIV RNA <400 c/mL at Baseline
Description: Virologic rebound was measured from the first dose of study therapy to the first of the 2 consecutive measurements ≥400 c/mL. Time to virologic rebound was analyzed using life tables. Measured Values show the Kaplan-Meier cumulative proportion of participants without virologic rebound up to the end of the respective interval.
Time Frame: Weeks 8-12, Weeks 20-24, Weeks 32-36, Weeks 44-48, Weeks 56-60, Weeks 68-72, Weeks 80-84, Weeks 92-96
Population: Treated subjects with HIV RNA <400 c/mL at baseline.
Measure: Number; unit: Proportion of participants
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 127 | 69
Proportion of participants
  By Weeks 8-12 | 0.9837 [0.31 to 22.68] | 1.000
  By Weeks 20-24 | 0.9837 [0.30 to 3.72] | 1.000
  By Weeks 32-36 | 0.9753 | 0.9841
  By Weeks 44-48 | 0.9669 | 0.9841
  By Weeks 56-60 | 0.9585 | 0.9841
  By Weeks 68-72 | 0.9585 | 0.9841
  By Weeks 80-84 | 0.9585 | 0.9674
  By Weeks 92-96 | 0.9585 | 0.9309
Statistical Analysis 1: Comparison: ATV/RTV Switch Arm vs PI/RTV Control Arm; Test type: Superiority or Other; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.3 to 3.72]

18. Secondary Outcome: Mean Change From Baseline in CD4 Count
Description: Mean change from baseline in CD4 count among treated subjects
Time Frame: Baseline, Week 48, Week 96
Population: Observed Cases (OC)
Measure: Mean (Standard Error); unit: cells/mm3
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Number analyzed (Participants) | 131 | 68
cells/mm3
  Week 48 (n=114; n=56) | 14 (13.1) | 44 (19.4)
  Week 96 (n=96; n=54) | 3 (16.9) | 82 (22.0)

ADVERSE EVENTS:
Arm/Group | ATV/RTV Switch Arm | PI/RTV Control Arm
Serious Adverse Events (participants affected / at risk) | 11/131 | 5/69
Other Adverse Events (participants affected / at risk) | 94/131 | 35/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATV/RTV Switch Arm (N=131) | PI/RTV Control Arm (N=69)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
DRUG ABUSE (Psychiatric disorders) | 1 | 0
DRUG DEPENDENCE (Psychiatric disorders) | 1 | 0
JAUNDICE (Hepatobiliary disorders) | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 3 | 0
PARALYSIS (Nervous system disorders) | 1 | 0
CONVULSION (Nervous system disorders) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0
NEUROSYPHILIS (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
CALCULUS BLADDER (Renal and urinary disorders) | 0 | 1
STEVENS-JOHNSON SYNDROME (Skin and subcutaneous tissue disorders) | 1 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 0
JAW FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
DRUG TOXICITY (Injury, poisoning and procedural complications) | 1 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATV/RTV Switch Arm (N=131) | PI/RTV Control Arm (N=69)
BLOOD BILIRUBIN INCREASED (Investigations) | 10 | 2
JAUNDICE (Hepatobiliary disorders) | 35 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 38 | 1
HEADACHE (Nervous system disorders) | 10 | 3
DIARRHOEA (Gastrointestinal disorders) | 10 | 5
INFLUENZA (Infections and infestations) | 10 | 1
SINUSITIS (Infections and infestations) | 5 | 4
BRONCHITIS (Infections and infestations) | 14 | 4
PHARYNGITIS (Infections and infestations) | 7 | 0
NASOPHARYNGITIS (Infections and infestations) | 8 | 2
URINARY TRACT INFECTION (Infections and infestations) | 4 | 5
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 13 | 13
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 11 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.